CLINICAL TRIAL: NCT03263481
Title: Intraductal Secretin Stimulation Test: What Is the Proper Collection Time?
Acronym: IDST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Evan Fogel, Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1203008365
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ERCP with inadvertent pancreatic cannulation (Experimental): Subjects undergoing ERCP for a biliary indication in which inadvertent pancreatic cannulation occurs will undergo intraductal secretin testing per the study protocol.
  Interventions: Procedure: Intraductal secretin test (IDST)

INTERVENTIONS:
Procedure: Intraductal secretin test (IDST) — If pancreatic duct entry incidentally occurs during the clinically scheduled ERCP and the pancreatic duct appears normal, an IDST will be performed for study purposes. An IDST consists of the administration of human secretin, after which pancreatic juice is collected intraductally. In this study, the fluid will be collected through continuous aspiration in 5 minute intervals for 30 minutes. Samples will be collected at 5, 10, 15, 20, 25, and 30 minutes after secretin administration (6 collections in total).

SUMMARY:
The aim is to evaluate the peak secretory flow rates and bicarbonate concentrations as determined by a 30 minute intraductal secretin stimulation test in patients with a low likelihood of pancreatic pathology and to compare these data to those obtained from our historical patients with suspected chronic pancreatitis. These will be patients in which inadvertent pancreatic cannulation occurs during therapeutic endoscopic retrograde cholangiopancreatography (ERCP) for biliary indications . All study subjects will receive a 5 day follow-up phone call. Enrollment goal is 36 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age referred to Indiana University Health, University Hospital for ERCP for a biliary indication, at the discretion of the treating MD (e.g. suspected common bile duct stone, initial post-liver transplant evaluation, suspected or confirmed cholangiocarcinoma, suspected primary sclerosing cholangitis -- see exclusion criterion #12)

Exclusion Criteria:

1. Pregnant woman or breast feeding
2. Age <18 years
3. Patient unable to give informed consent
4. Patient with a history of pancreatic surgery
5. Patient with a history of pancreatic cancer
6. Patient with a history of acute or chronic pancreatitis
7. Patient with radiographic evidence of acute or chronic pancreatitis on CT, MRCP, or EUS
8. Patient with a current or prior history of average daily alcohol consumption of greater than 60 g per day for more than 2 years
9. Patient with a history of cigarette smoking greater that 20 pack-years
10. Patient with a history of pancreas divisum
11. Evidence of chronic pancreatitis on pancreatogram during ERCP
12. ERCP for an isolated biliary indication with previous biliary sphincterotomy or for biliary stent exchange, when pancreatic entry should easily be avoided by the endoscopist.
13. History of allergy or adverse reactions to secretin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Secretory flow rates measured by volume | 5 minutes
  Volume of pancreatic juices will be collected
Secretory flow rates measured by volume | 10 minutes
  Volume of pancreatic juices will be collected
Secretory flow rates measured by volume | 15 minutes
  Volume of pancreatic juices will be collected
Secretory flow rates measured by volume | 20 minutes
  Volume of pancreatic juices will be collected
Secretory flow rates measured by volume | 25 minutes
  Volume of pancreatic juices will be collected
Secretory flow rates measured by volume | 30 minutes
  Volume of pancreatic juices will be collected
Bicarbonate concentration of timed pancreatic juice | 5 minutes
  Concentration of bicarbonate levels will be determined
Bicarbonate concentration of timed pancreatic juice | 10 minutes
  Concentration of bicarbonate levels will be determined
Bicarbonate concentration of timed pancreatic juice | 15 minutes
  Concentration of bicarbonate levels will be determined
Bicarbonate concentration of timed pancreatic juice | 20 minutes
  Concentration of bicarbonate levels will be determined
Bicarbonate concentration of timed pancreatic juice | 25 minutes
  Concentration of bicarbonate levels will be determined
Bicarbonate concentration of timed pancreatic juice | 30 minutes
  Concentration of bicarbonate levels will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Evan L Fogel, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States